CLINICAL TRIAL: NCT00554138
Title: Rosuvastatin Augments Dipyridamole Induced Vasodilation by Increased Adenosine Receptor Stimulation.
Brief Title: The Effect of Rosuvastatin on Adenosine Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: G.A. Rongen, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Rosudip01
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Adenosine Metabolism
Keywords: rosuvastatin; dipyridamole; caffeine
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental)
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: placebo — 1 dd for 7-10 days
  Arms: 1
Drug: rosuvastatin — 1 dd 20 mg for 7-10 days
  Arms: 2

SUMMARY:
The aim of this study is to show whether rosuvastatin influences adenosine metabolism. Therefore we will determine whether rosuvasatin increases dipyridamole-induced vasodilation by increased adenosine receptor stimulation.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 50 years
* Signed informed consent

Exclusion Criteria:

* hypertension
* hypercholesterolemia
* diabetes Mellitus
* alanine aminotransferase > 90 U/L
* creatinine Kinase > 440 U/L
* cardiovascular disease
* GFR < 80 ml/min

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
forearm vasodilatory response to dipyridamole | 7 days

SECONDARY OUTCOMES:
lipid profile | 7-10 days

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD, PhD, Study Director — Radboud University Medical Centre Dep. Pharmacology-Toxicology
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Meijer P, Oyen WJ, Dekker D, van den Broek PH, Wouters CW, Boerman OC, Scheffer GJ, Smits P, Rongen GA. Rosuvastatin increases extracellular adenosine formation in humans in vivo: a new perspective on cardiovascular protection. Arterioscler Thromb Vasc Biol. 2009 Jun;29(6):963-8. doi: 10.1161/ATVBAHA.108.179622. Epub 2009 Apr 9. PMID 19359665